CLINICAL TRIAL: NCT05362383
Title: Use of Transcutaneous Electrical Nerve Stimulation (TENS) for the Recovery of Oral Function After Orthognathic Surgery
Brief Title: Use of TENS for the Recovery of Oral Function After Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Alberto Cacho Casado, Associate Professor and Department Chair, Department of Dental Clinical Specialties, Faculty of Odontology, Complutense University, Madrid, Spain, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.P. - C.I. 12/136-E
Record Dates: First submitted 2022-04-24; First posted 2022-05-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Orthognathic Surgery; Physiology; Transcutaneous Electric Nerve Stimulation
Keywords: oral function
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): transcutaneous electrical nerve stimulation (TENS) is applied
  Interventions: Device: transcutaneous electrical nerve stimulation (TENS):Enraf Nonius® S82 model
- Control group (No Intervention): no intervention

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation (TENS):Enraf Nonius® S82 model — Will be used TENS device with a maximum frequency of 120 Hz and an intensity range of 0 to 99.5 milliampere. TENS electrodes (diameter 35-52 mm) will be placed bilaterally on mandibular elevator muscles, on the superficial masseter muscle above the gonial angle, and bilaterally on the anterior temporal muscle. The device will be applied in an identical manner to all patients in both groups and kept in position for the same time period (30 min) and for the control group the the device will be not switched on
  Arms: Experimental group

SUMMARY:
Oral functions of patients are markedly diminished immediately after orthognathic surgery, and novel approaches are needed to accelerate their recovery. The aim of this study is to examine the usefulness of weekly applications of transcutaneous electrical nerve stimulation (TENS) for this purpose, based on evidence of its effectiveness in other types of patients with muscle alterations. The main objective is to determine whether weekly TENS applications can increase the bite force and jaw opening in patients undergoing orthognathic surgery and decrease their pain and inflammation

DETAILED DESCRIPTION:
A single-blind randomized clinical trial will be conducted in patients scheduled for orthognathic surgery, divided between experimental and control groups. Participants will be selected by non-probabilistic sampling of consecutive patients until the estimated sample size is reached. All patients have a skeletal and facial deformity amenable to surgery after a pre-surgical orthodontic period. Patients will be randomly assigned to the experimental group for TENS application or the control group for sham-TENS and the researcher responsible for data analyses will be blinded also. Four variables will be measured: Maximum Jaw Opening using a digital dental caliber, Bite force measured using Dental Prescale Fuji® film, Pain using a visual analog scale (VAS) and facial inflammation using a soft ruler adapted to the contour of the patient's face. Data will be gathered from all patients on jaw opening, bite force, inflammation, and pain before surgery and at 7, 14, 21, and 28 days post-surgery, conducting measurements both before and after the TENS/sham-TENS session. TENS will be applied in an identical manner to all patients in both groups and kept in position for the same time period (30 min); however, the device will be not switched on for the control group, and the stimulation intensity will be adjusted for those in the experimental group to the maximum that did not cause discomfort or areas of contraction, maintaining this stimulation intensity and frequency throughout the 30-min session. Each participant will submit to a weekly TENS a weekly TENS or sham-TENS session on the same day of the week during a four-week period

ELIGIBILITY:
Inclusion Criteria:

* programing of bimaxillary or mandibular orthognathic surgery
* no previous or concomitant surgery for temporo-mandibular disorders
* no presence of complex syndromes
* no presence of muscle or nervous disorders or receipt of medication for such disorders

Exclusion Criteria:

* impossibility to attend follow-up appointments
* refusal of informed consent

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Bite force | Measurements will be taken baseline (before surgery)
  Bite force will be measured using Dental Prescale Fuji® film placed between the occlusal surfaces of the two arches, and the patient will be asked to bite as strongly as possible for 5 sec and the best-defined tooth print will be photographed with a Canon® EOS 500 camera (RAW format, F32, and annular Flash) at the minimum distance permitted by the 75-macro lens. The image will be processed in a Mac computer to obtain the color value according to the Cie L*a*b* (CIELAB) scale, which gives the color a numerical value.The corresponding pressure units (Megapascals, MPa) will be calculated according to Dental Prescale specifications, and the bite force (in Newtons [N]) will be obtained by using the following formula:
  Bite Force= Bite Pressure (MPa) x mm2 print surface.
Bite force | Measurements will be taken at 7 days after surgery
  Bite force will be measured using Dental Prescale Fuji® film placed between the occlusal surfaces of the two arches, and the patient will be asked to bite as strongly as possible for 5 sec and the best-defined tooth print will be photographed with a Canon® EOS 500 camera (RAW format, F32, and annular Flash) at the minimum distance permitted by the 75-macro lens. The image will be processed in a Mac computer to obtain the color value according to the Cie L*a*b* (CIELAB) scale, which gives the color a numerical value.The corresponding pressure units (Megapascals, MPa) will be calculated according to Dental Prescale specifications, and the bite force (in Newtons [N]) will be obtained by using the following formula:
  Bite Force= Bite Pressure (MPa) x mm2 print surface.
Bite force | Measurements will be taken at 14 days after surgery
  Bite force will be measured using Dental Prescale Fuji® film placed between the occlusal surfaces of the two arches, and the patient will be asked to bite as strongly as possible for 5 sec and the best-defined tooth print will be photographed with a Canon® EOS 500 camera (RAW format, F32, and annular Flash) at the minimum distance permitted by the 75-macro lens. The image will be processed in a Mac computer to obtain the color value according to the Cie L*a*b* (CIELAB) scale, which gives the color a numerical value.The corresponding pressure units (Megapascals, MPa) will be calculated according to Dental Prescale specifications, and the bite force (in Newtons [N]) will be obtained by using the following formula:
  Bite Force= Bite Pressure (MPa) x mm2 print surface.
Bite force | Measurements will be taken at 21 days after surgery
  Bite force will be measured using Dental Prescale Fuji® film placed between the occlusal surfaces of the two arches, and the patient will be asked to bite as strongly as possible for 5 sec and the best-defined tooth print will be photographed with a Canon® EOS 500 camera (RAW format, F32, and annular Flash) at the minimum distance permitted by the 75-macro lens. The image will be processed in a Mac computer to obtain the color value according to the Cie L*a*b* (CIELAB) scale, which gives the color a numerical value.The corresponding pressure units (Megapascals, MPa) will be calculated according to Dental Prescale specifications, and the bite force (in Newtons [N]) will be obtained by using the following formula:
  Bite Force= Bite Pressure (MPa) x mm2 print surface.
Bite force | Measurements will be taken at 28 days after surgery
  Bite force will be measured using Dental Prescale Fuji® film placed between the occlusal surfaces of the two arches, and the patient will be asked to bite as strongly as possible for 5 sec and the best-defined tooth print will be photographed with a Canon® EOS 500 camera (RAW format, F32, and annular Flash) at the minimum distance permitted by the 75-macro lens. The image will be processed in a Mac computer to obtain the color value according to the Cie L*a*b* (CIELAB) scale, which gives the color a numerical value.The corresponding pressure units (Megapascals, MPa) will be calculated according to Dental Prescale specifications, and the bite force (in Newtons [N]) will be obtained by using the following formula:
  Bite Force= Bite Pressure (MPa) x mm2 print surface.
Jaw opening | Measurements will be taken baseline (before surgery)
  Jaw opening will be evaluated with patients seated vertically upright in the dental chair, using a digital dental caliber (Model R 100110, Mestra®) to measure the maximum opening from the incisal margin of upper central incisors to the incisal margin of lower incisors, adding the amount (in mm) of overbite or subtracting the amount (in mm) of open bite in occlusion.
Jaw opening | Measurements will be taken at 7 days after surgery
  Jaw opening will be evaluated with patients seated vertically upright in the dental chair, using a digital dental caliber (Model R 100110, Mestra®) to measure the maximum opening from the incisal margin of upper central incisors to the incisal margin of lower incisors, adding the amount (in mm) of overbite or subtracting the amount (in mm) of open bite in occlusion.
Jaw opening | Measurements will be taken at 14 days after surgery
  Jaw opening will be evaluated with patients seated vertically upright in the dental chair, using a digital dental caliber (Model R 100110, Mestra®) to measure the maximum opening from the incisal margin of upper central incisors to the incisal margin of lower incisors, adding the amount (in mm) of overbite or subtracting the amount (in mm) of open bite in occlusion.
Jaw opening | Measurements will be taken at 21 days after surgery
  Jaw opening will be evaluated with patients seated vertically upright in the dental chair, using a digital dental caliber (Model R 100110, Mestra®) to measure the maximum opening from the incisal margin of upper central incisors to the incisal margin of lower incisors, adding the amount (in mm) of overbite or subtracting the amount (in mm) of open bite in occlusion.
Jaw opening | Measurements will be taken at 28 days after surgery
  Jaw opening will be evaluated with patients seated vertically upright in the dental chair, using a digital dental caliber (Model R 100110, Mestra®) to measure the maximum opening from the incisal margin of upper central incisors to the incisal margin of lower incisors, adding the amount (in mm) of overbite or subtracting the amount (in mm) of open bite in occlusion.
Pain (VAS) | Measurements will be taken baseline (before surgery)
  Pain perceived by patients while autonomously opening and closing their jaws will be evaluated using a visual analog scale (VAS) from 0 (least pain value) to 10 (value of greater pain).
Pain (VAS) | Measurements will be taken at 7 days after surgery
  Pain perceived by patients while autonomously opening and closing their jaws will be evaluated using a visual analog scale (VAS) from 0 (least pain value) to 10 (value of greater pain).
Pain (VAS) | Measurements will be taken at 14 days after surgery
  Pain perceived by patients while autonomously opening and closing their jaws will be evaluated using a visual analog scale (VAS) from 0 (least pain value) to 10 (value of greater pain).
Pain (VAS) | Measurements will be taken at 21 days after surgery
  Pain perceived by patients while autonomously opening and closing their jaws will be evaluated using a visual analog scale (VAS) from 0 (least pain value) to 10 (value of greater pain).
Pain (VAS) | Measurements will be taken at 28 days after surgery
  Pain perceived by patients while autonomously opening and closing their jaws will be evaluated using a visual analog scale (VAS) from 0 (least pain value) to 10 (value of greater pain).
Inflammation | Measurements will be taken baseline (before surgery)
  Inflammation will be measured (in mm) with patients seated upright in the dental chair, using a soft ruler to obtain a horizontal measurement from the lower border of the earlobe to the corner of the mouth and a vertical measurement from the gonial angle to the outer canthus of the eye. The soft ruler will be adapted to the contour of the patient's face without exerting any pressure.
Inflammation | Measurements will be taken at 7 days after surgery
  Inflammation will be measured (in mm) with patients seated upright in the dental chair, using a soft ruler to obtain a horizontal measurement from the lower border of the earlobe to the corner of the mouth and a vertical measurement from the gonial angle to the outer canthus of the eye. The soft ruler will be adapted to the contour of the patient's face without exerting any pressure.
Inflammation | Measurements will be taken at 14 days after surgery
  Inflammation will be measured (in mm) with patients seated upright in the dental chair, using a soft ruler to obtain a horizontal measurement from the lower border of the earlobe to the corner of the mouth and a vertical measurement from the gonial angle to the outer canthus of the eye. The soft ruler will be adapted to the contour of the patient's face without exerting any pressure.
Inflammation | Measurements will be taken at 21 days after surgery
  Inflammation will be measured (in mm) with patients seated upright in the dental chair, using a soft ruler to obtain a horizontal measurement from the lower border of the earlobe to the corner of the mouth and a vertical measurement from the gonial angle to the outer canthus of the eye. The soft ruler will be adapted to the contour of the patient's face without exerting any pressure.
Inflammation | Measurements will be taken at 28 days after surgery
  Inflammation will be measured (in mm) with patients seated upright in the dental chair, using a soft ruler to obtain a horizontal measurement from the lower border of the earlobe to the corner of the mouth and a vertical measurement from the gonial angle to the outer canthus of the eye. The soft ruler will be adapted to the contour of the patient's face without exerting any pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto C Cacho, Prof, Principal Investigator — Faculty of Odontology, University Complutense, Madrid
Locations (1):
- Faculty of Odontology, University Complutense, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teng TT, Ko EW, Huang CS, Chen YR. The Effect of early physiotherapy on the recovery of mandibular function after orthognathic surgery for Class III correction: part I--jaw-motion analysis. J Craniomaxillofac Surg. 2015 Jan;43(1):131-7. doi: 10.1016/j.jcms.2014.10.025. Epub 2014 Nov 1. PMID 25439086
- [Background] Wen-Ching Ko E, Huang CS, Lo LJ, Chen YR. Longitudinal observation of mandibular motion pattern in patients with skeletal Class III malocclusion subsequent to orthognathic surgery. J Oral Maxillofac Surg. 2012 Feb;70(2):e158-68. doi: 10.1016/j.joms.2011.10.002. PMID 22260918
- [Background] Jung HD, Jung YS, Park JH, Park HS. Recovery pattern of mandibular movement by active physical therapy after bilateral transoral vertical ramus osteotomy. J Oral Maxillofac Surg. 2012 Jul;70(7):e431-7. doi: 10.1016/j.joms.2012.02.033. PMID 22698299
- [Background] Bell WH, Gonyea W, Finn RA, Storum KA, Johnston C, Throckmorton GS. Muscular rehabilitation after orthognathic surgery. Oral Surg Oral Med Oral Pathol. 1983 Sep;56(3):229-35. doi: 10.1016/0030-4220(83)90001-4. PMID 6579456
- [Background] Oh DW, Kim KS, Lee GW. The effect of physiotherapy on post-temporomandibular joint surgery patients. J Oral Rehabil. 2002 May;29(5):441-6. doi: 10.1046/j.1365-2842.2002.00850.x. PMID 12028491
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Sato KL, Sanada LS, Rakel BA, Sluka KA. Increasing intensity of TENS prevents analgesic tolerance in rats. J Pain. 2012 Sep;13(9):884-90. doi: 10.1016/j.jpain.2012.06.004. Epub 2012 Aug 1. PMID 22858165
- [Background] Dowswell T, Bedwell C, Lavender T, Neilson JP. Transcutaneous electrical nerve stimulation (TENS) for pain relief in labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007214. doi: 10.1002/14651858.CD007214.pub2. PMID 19370680
- [Background] Tong KC, Lo SK, Cheing GL. Alternating frequencies of transcutaneous electric nerve stimulation: does it produce greater analgesic effects on mechanical and thermal pain thresholds? Arch Phys Med Rehabil. 2007 Oct;88(10):1344-9. doi: 10.1016/j.apmr.2007.07.017. PMID 17908580
- [Background] Liebano RE, Rakel B, Vance CGT, Walsh DM, Sluka KA. An investigation of the development of analgesic tolerance to TENS in humans. Pain. 2011 Feb;152(2):335-342. doi: 10.1016/j.pain.2010.10.040. Epub 2010 Dec 8. PMID 21144659
- [Background] Mendell LM. Constructing and deconstructing the gate theory of pain. Pain. 2014 Feb;155(2):210-216. doi: 10.1016/j.pain.2013.12.010. Epub 2013 Dec 12. PMID 24334188
- [Background] Iwase M, Ohashi M, Tachibana H, Toyoshima T, Nagumo M. Bite force, occlusal contact area and masticatory efficiency before and after orthognathic surgical correction of mandibular prognathism. Int J Oral Maxillofac Surg. 2006 Dec;35(12):1102-7. doi: 10.1016/j.ijom.2006.08.014. Epub 2006 Nov 9. PMID 17097270
- [Background] Hidaka O, Iwasaki M, Saito M, Morimoto T. Influence of clenching intensity on bite force balance, occlusal contact area, and average bite pressure. J Dent Res. 1999 Jul;78(7):1336-44. doi: 10.1177/00220345990780070801. PMID 10403461
- [Background] Matsui Y, Ohno K, Michi K, Suzuki Y, Yamagata K. A computerized method for evaluating balance of occlusal load. J Oral Rehabil. 1996 Aug;23(8):530-5. doi: 10.1111/j.1365-2842.1996.tb00891.x. PMID 8866265
- [Background] Ohkura K, Harada K, Morishima S, Enomoto S. Changes in bite force and occlusal contact area after orthognathic surgery for correction of mandibular prognathism. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Feb;91(2):141-5. doi: 10.1067/moe.2001.112334. PMID 11174588
- [Background] Yaedu RYF, Mello MAB, Tucunduva RA, da Silveira JSZ, Takahashi MPMS, Valente ACB. Postoperative Orthognathic Surgery Edema Assessment With and Without Manual Lymphatic Drainage. J Craniofac Surg. 2017 Oct;28(7):1816-1820. doi: 10.1097/SCS.0000000000003850. PMID 28872503
- [Background] Moran F, Leonard T, Hawthorne S, Hughes CM, McCrum-Gardner E, Johnson MI, Rakel BA, Sluka KA, Walsh DM. Hypoalgesia in response to transcutaneous electrical nerve stimulation (TENS) depends on stimulation intensity. J Pain. 2011 Aug;12(8):929-35. doi: 10.1016/j.jpain.2011.02.352. Epub 2011 Apr 9. PMID 21481649
- [Background] Throckmorton GS, Ellis E 3rd, Buschang PH. Morphologic and biomechanical correlates with maximum bite forces in orthognathic surgery patients. J Oral Maxillofac Surg. 2000 May;58(5):515-24. doi: 10.1016/s0278-2391(00)90014-4. PMID 10800907
- [Background] Trawitzki LV, Silva JB, Regalo SC, Mello-Filho FV. Effect of class II and class III dentofacial deformities under orthodontic treatment on maximal isometric bite force. Arch Oral Biol. 2011 Oct;56(10):972-6. doi: 10.1016/j.archoralbio.2011.02.018. Epub 2011 Mar 25. PMID 21440242
- [Background] Nagai I, Tanaka N, Noguchi M, Suda Y, Sonoda T, Kohama G. Changes in occlusal state of patients with mandibular prognathism after orthognathic surgery: a pilot study. Br J Oral Maxillofac Surg. 2001 Dec;39(6):429-33. doi: 10.1054/bjom.2001.0681. PMID 11735137
- [Background] Ueki K, Marukawa K, Hashiba Y, Nakagawa K, Degerliyurt K, Yamamoto E. Assessment of the relationship between the recovery of maximum mandibular opening and the maxillomandibular fixation period after orthognathic surgery. J Oral Maxillofac Surg. 2008 Mar;66(3):486-91. doi: 10.1016/j.joms.2007.08.044. PMID 18280381
- [Background] Oliveira Sierra S, Melo Deana A, Mesquita Ferrari RA, Maia Albarello P, Bussadori SK, Santos Fernandes KP. Effect of low-level laser therapy on the post-surgical inflammatory process after third molar removal: study protocol for a double-blind randomized controlled trial. Trials. 2013 Nov 6;14:373. doi: 10.1186/1745-6215-14-373. PMID 24195796
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT05362383/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT05362383/SAP_001.pdf